CLINICAL TRIAL: NCT05121714
Title: A Two Part, Fixed-sequence, Open-label Crossover Study to Evaluate Potential CYP1A2-mediated Drug-drug Interactions of ABX464 in Healthy Subjects Using Caffeine and Fluvoxamine as Probe Drugs
Brief Title: Evaluation of the Potential CYP1A2-mediated Drug Drug Interaction Safety, and Tolerability of ABX464
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abivax S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ABX464-902
Record Dates: First submitted 2021-10-11; First posted 2021-11-16 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Healthy
MeSH Terms: interventions — Caffeine; ABX464; Fluvoxamine

STUDY DESIGN:
Intervention Model Description: This is a Phase 1, 2 part, fixed-sequence open-label, crossover study to evaluate the potential CYP1A2-mediated drug-drug interactions (DDI), safety, and tolerability of ABX464 combined with a known CYP1A2 substrate (caffeine) and a known CYP1A2 inhibitor (fluvoxamine). Sixty (60) healthy adult male and female subjects 18 to 55 years of age are planned to participate in the study. Separate cohorts of subjects will be enrolled for Part A (24 subjects) and Part B (36 subjects).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Evaluation of CYP1A2 inhibition and induction potential by ABX464 (Other): Using a fixed-sequence crossover study design, the Pharmacokinetics (PK) of caffeine (50 milligrams (mg) single oral dose) will be evaluated in the absence and presence of ABX464 (50 mg once daily for 14 days) in 24 healthy subjects. Caffeine will be administered on Day 1 in the absence of ABX464, on Day 4 simultaneously with ABX464 to evaluate potential CYP1A2 inhibition by ABX464, and on Day 17 simultaneously with ABX464 following 14 days of once daily dosing of ABX464 to evaluate potential CYP1A2 induction by ABX464.
  Interventions: Drug: Caffeine; Drug: ABX464
- Evaluation of ABX464 as a substrate for CYP1A2 (Other): Using a fixed-sequence crossover study design, the PK of ABX464 (50 mg single oral dose) will be evaluated in the absence and presence of fluvoxamine (100 mg once daily for 10 days) in 36 healthy subjects. ABX464 will be administered on Day 1 in the absence of fluvoxamine and on Day 11 simultaneously with fluvoxamine following 10 days of once daily dosing of fluvoxamine to evaluate whether ABX464 is a substrate for CYP1A2
  Interventions: Drug: ABX464; Drug: Fluvoxamine

INTERVENTIONS:
Drug: Caffeine — This is a 2 part, fixed-sequence open-label, crossover study to evaluate the potential CYP1A2-mediated drug-drug interactions (DDI), safety, and tolerability of ABX464 combined with a known CYP1A2 substrate (caffeine)
  Arms: Evaluation of CYP1A2 inhibition and induction potential by ABX464
Drug: ABX464 — This is a 2 part, fixed-sequence open-label, crossover study to evaluate the potential CYP1A2-mediated drug-drug interactions (DDI), safety, and tolerability of ABX464 combined with a known CYP1A2 inhibitor (fluvoxamine) and a known CYP1A2 substrate (caffeine).
Drug: Fluvoxamine — his is a 2 part, fixed-sequence open-label, crossover study to evaluate the potential CYP1A2-mediated drug-drug interactions (DDI), safety, and tolerability of ABX464 combined with a known CYP1A2 inhibitor (fluvoxamine).
  Arms: Evaluation of ABX464 as a substrate for CYP1A2

SUMMARY:
A two part, fixed-sequence, open-label crossover study to evaluate potential CYP1A2-mediated drug-drug interactions of ABX464 in healthy subjects using caffeine and fluvoxamine as probe drugs

DETAILED DESCRIPTION:
This is a Phase 1, 2 part, fixed-sequence open-label, crossover study to evaluate the potential CYP1A2-mediated drug-drug interactions (DDI), safety, and tolerability of ABX464 combined with a known CYP1A2 substrate (caffeine) and a known CYP1A2 inhibitor (fluvoxamine). Sixty (60) healthy adult male and female subjects 18 to 55 years of age are planned to participate in the study. Separate cohorts of subjects will be enrolled for Part A (24 subjects) and Part B (36 subjects).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, male or female subject, between 18 and 55 years of age, inclusive.
2. Women of childbearing potential (WOCBP) and men receiving the study treatment and their partners must agree to use a highly effective contraceptive method during the study and for 6 months (180 days) after end of study or early termination.
3. Subject with a body mass index (BMI) of 18.5-30 kilogrammes per square metre (kg/m²).
4. No clinically significant history of previous allergy / sensitivity to ABX464 or any of the excipients within the IMP.
5. No clinically significant history of previous allergy / sensitivity to caffeine (for Part A) or fluvoxamine (for Part B), or any of the excipients contained within the Non-Investigational Medicinal Product (NIMP).
6. No clinically significant abnormal test results for serum biochemistry, haematology and/or urine analyses within 28 days before the first dose administration of the Investigational Medicinal Product (IMP)/NIMP.
7. Subject with a negative urinary drugs of abuse (DOA) screen (including alcohol and cotinine) test results, determined within 28 days before the first dose administration of the IMP (N.B.: A positive result may be repeated at the Investigator's discretion).
8. Subject with negative human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg)) and hepatitis C virus antibody (HCV Ab) results at Screening.
9. No known history of hypertension or abnormal vital signs at screening defined as supine systolic blood pressure (SBP) < 90 or > 140 millimetres of mercury (mmHg), and pulse rate < 40 or > 90 beats per minute (bpm).
10. No clinically significant abnormalities in 12-lead electrocardiogram (ECG) determined within 28 days before first dose of IMP including PR > 220 milliseconds (ms) and QT interval corrected using Fridericia formula (QTcF) >450 ms in males or >470 ms in females, or evidence of clinically significant dysrhythmias (long QT features on ECG, left bundle branch block, or ventricular arrhythmia), atrial fibrillation or history of familial long QT syndromes (Note: partial right bundle branch block is acceptable).
11. Subject must be available to complete the study (including all follow up visits/phone call).
12. Subject must satisfy an Investigator about their fitness to participate in the study.
13. Subject must provide written informed consent to participate in the study

Exclusion Criteria:

1. Female subject who is pregnant, currently lactating or breastfeeding.
2. A clinically significant history of gastrointestinal disorder likely to influence IMP absorption.
3. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements, or any product known to interact with CYP1A2 within 28 days or 5 half-lives (whichever is longer) prior to the first dose of IMP.
4. Subject who has, or who have a relevant history of any clinically significant: neurological, gastrointestinal, renal, hepatic, cardiovascular, vascular, psychiatric, respiratory, metabolic, endocrine, or haematological conditions and/or other significant medical conditions including, without limitation, those pertaining to coronavirus disease 2019 (COVID-19) that, in the opinion of the Investigator or their appropriately qualified designee, would jeopardise the safety of the subject, safety of anyone involved in the study or impact on the validity of the study results.
5. A clinically significant history of drug or alcohol abuse (defined as the consumption of more than 14 units for male and female subjects) of alcohol a week) within the past two years.
6. Inability to communicate well with the Investigators (i.e., language problem, poor mental development or impaired cerebral function).
7. Participation in a New Chemical Entity (NCE) clinical study within 3 months or five half-lives, whichever is longer, or a marketed drug clinical study within 30 days or five half-lives, whichever is longer, before the first dose of IMP (Washout period between studies is defined as the period of time elapsed between the last dose of the previous study and the first dose of the next study).
8. Donation of 450 millilitres (mL) or more blood within the 3 months before the first dose of IMP.
9. Users of nicotine products i.e., current smokers or ex-smokers who have smoked within 6 months prior to first dose administration with the study medication or users of cigarette replacements (i.e., e-cigarettes, nicotine patches or gums).
10. Total serum bilirubin, alkaline phosphatase (ALP), aspartate transaminase (AST) / serum glutamic-oxaloacetic transaminase (SGOT) and alanine transaminase (ALT) / Serum glutamic pyruvic transaminase (SGPT) > 1.5 x upper limit of normal (ULN).
11. Experiences regular headaches (i.e., experiences headaches more than weekly).

    Part B Only:
12. Meets Diagnostic and Statistical Manual of Mental Disorders (5th Edition) criteria for moderate or severe substance use disorder within 6 months before Screening.
13. Reports having experienced suicidal ideation (Type 4 or 5 on the Columbia-Suicide Severity Rating Scale [C-SSRS]) within 30 days prior to Screening, any suicidal behaviour within 2 years prior to Screening (Any "Yes" answers on Suicidal Behaviour section of C-SSRS), and/or the Investigator assesses the subject to be a safety risk to him/herself or others;
14. Clinically significant history of depression or anxiety.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
Part A Evaluate the potential for inhibition and/or induction of CYP1A2 in vivo based on the Peak Plasma Concentration (Cmax) of caffeine (a known CYP1A2 substrate) in the presence and absence of ABX464. | Day 1, Day 4 and Day 17
  Peak Plasma Concentration (Cmax) for caffeine
Part A Evaluate the potential for inhibition and/or induction of CYP1A2 in vivo based on the Area under the plasma concentration versus time curve (AUC) of caffeine (a known CYP1A2 substrate) in the presence and absence of ABX464. | Day 1, Day 4 and Day 17
  Area under the plasma concentration versus time curve (AUC) for caffeine
Part B Evaluate whether ABX464 is a substrate for CYP1A2 in vivo based on Peak Plasma Concentration (Cmax) in the presence and absence of fluvoxamine. | Day 1 and Day11
  Peak Plasma Concentration (Cmax) for ABX464
Part B Evaluate whether ABX464 is a substrate for CYP1A2 in vivo based on Area under the plasma concentration versus time curve (AUC) in the presence and absence of fluvoxamine. | Day 1 and Day 11
  Area under the plasma concentration versus time curve (AUC) for ABX464

SECONDARY OUTCOMES:
Parts A & B • Evaluate the safety and tolerability of ABX464 alone and in the presence of caffeine or fluvoxamine | from baseline up to Day 25
  Incidence of Adverse Events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Gineste, Study Director — Abivax S.A.
Locations (1):
- Simbec-Orion, Merthyr Tydfil, United Kingdom

IPD SHARING:
Plan to Share IPD: No